CLINICAL TRIAL: NCT06801665
Title: Fecal Microbiota Transplantation Combined With QL1706, Bevacizumab, and XELOX as First-line Treatment for Advanced MSS-type Colon Cancer With Liver Metastasis: A Prospective, Multi-center, Single-arm Phase II Study
Brief Title: FMT+ QL1706+Bevacizumab+ XELOX as First-line Treatment for Advanced MSS-type Colon Cancer With Liver Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hua Jiang (Other)
Responsible Party: Sponsor-Investigator, Hua Jiang, Director, Changzhou No.2 People's Hospital
Organization: Changzhou No.2 People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2024]YLJSA162
Record Dates: First submitted 2025-01-25; First posted 2025-01-30 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Colon Cancer Liver Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT+QL1706+Bevacizumab+XELOX (Experimental)
  Interventions: Combination Product: FMT+QL1706+Bevacizumab+XELOX

INTERVENTIONS:
Combination Product: FMT+QL1706+Bevacizumab+XELOX — Participants will receive FMT combined with QL1706+Bevacizumab+XELOX for 6 cycles. If there is no progression of the disease after 6 cycles of the first-line treatment, then patients will enter the maintenance treatment stage. The therapy of maintenance treatment stage was at the discretion of the investigator.

SUMMARY:
The investigators plan to initiate a prospective, multicenter, phase II study, recruiting 30 patients with advanced colon cancer patients with liver metastasis who have not received prior treatment. This study plans to reconstruct intestinal microecology through fecal microbiota transplantation (FMT), and combine with QL1706+Bevacizumab+XELOX to enhance the anti-tumor immune effect at the same time, thereby improving the prognosis of colon cancer patients with liver metastasis.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-center, exploratory clinical study. Patients with previously untreated, newly diagnosed advanced colon cancer with liver metastasis, who could be diagnosed by histological or cytological means, ECOG PS 0-1, excluded Ras, Raf wild type left colon and rectum, excluded dMMR/MSI-H. Eligible subjects who met the inclusion criteria were screened and signed informed consent.

FMT was performed 2 days before treatment with QL1706, bevacizumab, and chemotherapy. QL1706， bevacizumab, and chemotherapy (XELOX) were administered every 3 weeks according to the patient's body surface area. A total of 6 cycles were performed. Subsequent maintenance therapy was at the discretion of the investigator.

RECIST v1.1 was used for tumor evaluation every 6 weeks during treatment. NCI-CTCAE 5.0 was used for safety assessment every 3 weeks. Adverse events were recorded throughout the study to 90 days after the end of treatment. Treatment continues until disease progression, subject withdraws informed consent, loss of follow-up, or death. Patients should provide 10ml whole blood samples and fecal samples at baseline, after two cycles of treatment, after four cycles of treatment, before maintenance treatment for the detection of efficacy prediction markers (each cycle is 21 days).

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmed advanced colon cancer with liver metastasis.
2. Signed written informed consent.
3. Have not received anti-tumor treatment.
4. According to the investigators assessment, at least one measurable target lesion defined by RECIST v1.1.
5. Patients of both sexes, aged ≥18 years and ≤75 years.
6. ECOG PS 0-1;
7. Expected survival time ≥ 3 months;
8. Have adequate organ and bone marrow function, laboratory examination within 7 days prior to enrollment meets the following requirements, as follows:

1) Blood routine: ANC ≥ 1.5 × 10^9/L, Platelet count ≥ 100 × 10^9/L, HGB ≥100 g/L (no blood transfusion or erythropoietin dependence within 14 days); 2) Liver function: TBIL ≤1.5 x ULN; ALT/AST ≤ 5 x ULN; ALP ≤5×ULN; 3) Renal function: Cr ≤1.5×ULN, or creatinine clearance ≥50 mL/min: Urine routine results showed urinary protein < 2+; 4) Coagulation function: INR or PT ≤1.5 x ULN. 9.For female subjects of reproductive age, a urine or serum pregnancy test should be performed and the result is negative 3 days prior to receiving the initial study drug administration.

10. For women of childbearing potential (WOCBP): agreement to refrain from heterosexual intercourse or use contraception.

11. For men: agreement to refrain from heterosexual intercourse or use a condom, and agreement to refrain from donating sperm.

Exclusion Criteria:

1. Suffered from other malignancies in the past 5 years, excluding cured basal cell carcinoma of the skin, cervical carcinoma in situ and papillary thyroid carcinoma.
2. Patients requiring elective surgery during the trial.
3. Patients who cannot take oral drugs, or have conditions that the investigator determines to significantly affect gastrointestinal absorption, such as chronic diarrhea, intestinal obstruction, etc., and are not suitable for treatment.
4. Patients during pregnancy (positive pregnancy test) or lactation.
5. Central nervous system metastasis or meningeal metastasis.
6. Uncontrollable bone metastasis, or patients at risk of fracture, requiring surgery, local radiation therapy.
7. Patients with active infection requiring systemic anti-infection treatment.
8. Patients with a history of immunodeficiency, including those who are positive for HIV antibody tests.
9. Patients with known, active autoimmune diseases.
10. Patients with uncontrolled active hepatitis B, patients with hepatitis C virus infection (HCV antibody positive).
11. A history of severe cardiovascular and cerebrovascular diseases, including but not limited to: severe arrhythmia, acute coronary syndrome within 6 months, congestive heart failure, aortic dissection, stroke, and T IA history.
12. Severe bleeding events occur within half a year, or high bleeding risk factors such as active digestive tract ulcers and esophageal and gastric varices due to liver cirrhosis.
13. Patients with diabetes who cannot be stably controlled by drugs (including insulin).
14. Mental or language disorders that prevent communication with the patient;
15. Patients participating in another clinical trial.
16. MSI-H/ d MMR without immunotherapy; left colorectum of Ras, Raf wild-type.
17. The investigator believes that the subject has other serious systemic diseases or other conditions that make him unsuitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months
  Objective response rate will be assessed by investigators.

SECONDARY OUTCOMES:
Median Progression-Free Survival (mPFS) | up to 24 months
  Observation for mPFS will be recorded until the end of follow-up after the start of 1st cycle of treatment.
Median Overall Survival (mOS) | up to 24 months
  The time from the first treatment to death from any cause.
6-Months Progression-Free Survival Rate (6month-PFS) | up to 6 months
  The proportion of patients whose disease did not progress 6 months after treatment
12-Months Progression-Free Survival Rate (12month-PFS) | up to 12 months
  The proportion of patients whose disease did not progress 12 months after treatment
18-Months Progression-Free Survival Rate (18month-PFS) | up to 18 months
  The proportion of patients whose disease did not progress 18 months after treatment
6-Months overall survival rate(6-Months-OS Rate) | up to 6 months
  The proportion of patients who have not died after 6-Months of treatment
12-Months overall survival rate(12-Months-OS Rate) | up to 12 months
  The proportion of patients whose disease did not progress 12 months after treatment
18-Months overall survival rate(18-Monthsr-OS Rate) | up to 18 months
  The proportion of patients who have not died after 18 months of treatment
Objective Response Rate (ORR) of liver metastases | up to 24 months
  Objective response rate will be assessed by investigators.
Disease Control Rate (DCR) | up to 24 months
  The proportion of patients whose tumors achieve a response (CR+PR) and stable disease (SD) after treatment for the minimum duration required.
Surgical conversion rate | up to 24 months
  Proportion of inoperable patients converted to operable.
Incidence of Adverse events (AEs) | up to 24 months
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).
Quality of Life (QoL) | up to 24 months
  QoL(quality of life) will be evaluated by EORTC-QLQ-C30.The total score ranges from 0 to 60, with higher scores indicating better quality of life
The Diversity of Fecal Microbiota | up to 24 months
  This will be detected by 16s rRNA sequencing or metagenomes.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second People's Hospital of Changzhou, Changzhou, China

IPD SHARING:
Plan to Share IPD: No